CLINICAL TRIAL: NCT00073203
Title: A 6- Week, Randomized, Double-Blind, Parallel-Group, Active-and Placebo-Controlled Trial to Assess the Efficacy of R228060 in Adult Subjects With Major Depressive Disorder (MDD)
Brief Title: A 6 Week Study to Determine the Effectiveness of R228060 in Adult Subjects With Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR004339
Record Dates: First submitted 2003-11-17; First posted 2003-11-19 (Estimated); Last update posted 2009-08-28 (Estimated); Status verified 2004-05

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Paroxetine

INTERVENTIONS:
Drug: R228060
Drug: Placebo and Paroxetine

SUMMARY:
The purpose of this research study is to determine the effectiveness of 2 target doses of R228060 in comparison with placebo during 6 weeks of treatment in moderately to severely depressed adult subjects with major depressive disorder.

Approximately 488 subjects will be involved in the study.

ELIGIBILITY:
* Generally healthy adults on the basis of a physical examination, medical history, ECG and laboratory work-up.
* Subject needs to meet criteria for diagnosis of moderate or severe major depression as defined by the protocol.
* The subject also needs to be an outpatient to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488
Dates: Study Completion 2004-05

CONTACTS AND LOCATIONS:
Locations (1):
- JJ PRD Research Center, Titusville, New Jersey, United States